CLINICAL TRIAL: NCT02919046
Title: Single Arm and Multicenter Clinical Trial to Evaluating the Efficacy and Safety of the Chimeric Antigen Receptor T Cell Immunotherapy (CAR-T) for Relapsed or Refractory Neuroblastoma in Children
Brief Title: Study Evaluating the Efficacy and Safety With CAR-T for Relapsed or Refractory Neuroblastoma in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sinobioway Cell Therapy Co., Ltd. (Industry)
Collaborators: Nanjing Children's Hospital (Other); Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WM-CART-07
Record Dates: First submitted 2016-09-26; First posted 2016-09-29 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Relapsed or Refractory Neuroblastoma
Keywords: neuroblastoma; CAR-T
MeSH Terms: conditions — Recurrence; Neuroblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm (Experimental): Name:The Chimeric Antigen Receptor T Cell Immunotherapy (CAR-T) Dosage form：injection Dosage:100ml/time Frequency:0 days,the first day,the second day,29 days,30 days Duration:Total five times
  Interventions: Biological: GD2-targeted CAR-T cells

INTERVENTIONS:
Biological: GD2-targeted CAR-T cells — This study have only one arm that is CAR-T experimental arm. Firstly all participators will be attended the screening, who passed the screening for the treatment of CAR-T cells, the CAR-GD2-modified T cells can recognize and kill tumor cells in the body，follow-up 35 months.

SUMMARY:
This single-arm, multicenter clinical study will treat the patient who have relapsed or refractory neuroblastoma with an infusion of the patient's own T cells that have been genetically modified to express a chimeric antigen receptor(CAR)that will bind to tumour cells modified to express the GD2 protein on the cell surface. The study will determine if these modified T cells help the body's immune system eliminate tumour cells .The trial will also study the safety of treatment for CAR-T, how long CAR-T cells stay in the patient's body and the impact on this treatment for survival.

DETAILED DESCRIPTION:
This is a single-arm, multicenter clinical study to evaluate efficacy and safety of chimeric antigen receptor T cell immunotherapy (CAR-T) in the treatment of relapsed or refractory neuroblastoma in children. The study will be conducted using a phaseⅠ/Ⅱdesign the study will have the following sequential phases: part A (screening, leukapheresis,cell product preparation and cytoreductive chemotherapy) and part B (treatment and follow-up). the follow-up period for each participant is approximately 35 months after the final CAR-T infusion. The total duration of the study are expected to be approximately 3 years. A total of 22 patients may be enrolled over a period of 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Up to diagnostic criteria for relapsed or refractory neuroblastoma or high-risk patients，including:

   * Relapsed neuroblastoma : Children diagnosed with neuroblastoma who after standard treatment and remission, present lesions again and cannot reach complete remission with surgery.
   * Refractory neuroblastoma : ① Untreated patients that do not have to reach completes remission after 4 courses of chemotherapy in accordance with standard regimens nor reach complete remission with surgery. ② High-risk patients : Who have cell genetic variation, such as MYCN amplification or bone marrow metastasis.
2. Relapsed or Refractory Neuroblastoma: Target, of which expression may be intervened , discovered with Immunohistochemistry can be selected (GD2 +) (more than 50% of tumor cells is at least 2+ , adopting anti-GD2-mAb14G2a ).
3. Age: 1~14 years old of age at the time of enrollment, male or female.
4. Physical condition is good: ECOG score reaches 0 to 2 points.
5. Body weights greater than or equal to 10 kg.
6. White blood cell counts acuity≥ 1.0 x10^9 / L.
7. Estimated survival times > 90 days.
8. Voluntary participation, good compliance, can cooperate with the experimental observation and signed an informed consent form.

Exclusion Criteria:

1. Positive pregnancy tests.
2. Uncontrolled infection.
3. HIV infection, hepatitis B or C activity period.
4. Patients who need long-term immunosuppressive therapy (Such as allergies, autoimmune diseases, GVHD, etc.)
5. Combined activity of the central nervous system malignant tumor invasion.
6. Abnormal coagulation function, patients with severe thrombosis.
7. Organ failure

   1. Heart：class Ⅱ or above.
   2. Liver：class Ⅱ or above( Refer to Classification of Wuhan Conference (1983)).
   3. Kidney: The second stage of renal insufficiency or above.
   4. Lung: class Ⅱdecreased slightly or above.
   5. Brain: The central nervous system transfer or have active lesions.
8. Patients who have participated in other clinical trials or other clinical trials in the past 30 days.
9. The researchers believe that the patient is not suitable to participate in the study.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2016-09; Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
The overall efficiency of patients with neuroblastoma after autologous CAR-T cell therapy | 28d,56d,90d
  The overall efficiency will be determined by the evaluation of CT/MRI scans and bone marrow biopsy. Assessment of tumor remission rate according to International Neuroblastoma Response Criteria. The overall efficiency = (complete remission (CR) number + the number of very good partial remission (VGPR) number + partial response (PR) number + mixed reaction (MR) number + no response (NR) number) / total number of cases receiving treatment.

SECONDARY OUTCOMES:
Progression free survival | 3 years
  From the test of the progression of disease progression or the interval between disease and death.
Overall survival | 3 years
  For all patients, overall survival refers to the period from being included in the test group to death caused by any reason
Patients-based Quality of Life Evaluation | 3 years
  According to EORTC quality of life measurement scale PedsQL4.0_ children's quality of life of the core scale of the evaluation and comparison of physical condition before and after treatment.
3°or above incidence rate of serious adverse reaction related to treatment | 3 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Fang, Ph.D, Principal Investigator — Nanjing Children's Hospital; Kuiran Dong, Ph.D, Principal Investigator — Children's Hospital of Fudan University
Locations (2):
- China (2):
  - Nanjing Children's Hospital, Nanjing, Jiangsu
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thomas S, Straathof K, Himoudi N, Anderson J, Pule M. An Optimized GD2-Targeting Retroviral Cassette for More Potent and Safer Cellular Therapy of Neuroblastoma and Other Cancers. PLoS One. 2016 Mar 31;11(3):e0152196. doi: 10.1371/journal.pone.0152196. eCollection 2016. PMID 27030986
- See also: An Optimized GD2-Targeting Retroviral Cassette for More Potent and Safer Cellular Therapy of Neuroblastoma and Other Cancers — http://dx.doi.org/10.1371/journal.pone.0152196